CLINICAL TRIAL: NCT00035516
Title: A Phase II Study of Epothilone Analog BMS-247550 in Patients With Non-Small Cell Lung Cancer Who Have Failed First Line Platinum Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Purpose: Treatment
Other Study IDs: CA163-011
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Carcinoma, Non-small-cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Epothilones

INTERVENTIONS:
Drug: Epothilone

SUMMARY:
The purpose of this clinical research study is to learn if BMS-247550 can shrink or slow the growth of the cancer in patients with non-small cell lung cancer who have failed first-line platinum based chemotherapy. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer
* Bidimensionally measurable disease
* Progressed following therapy with one prior cisplatin or carboplatin based chemotherapy regimen for Stage III or IV or metastatic recurrent disease
* Adequate hematologic function as defined by: absolute neutrophils =/> 2,000/mm3, and platelets > 125,000/mm3
* Adequate hepatic function as defined by: serum bilirubin=/<1.5 times the upper institutional limits of normal, ALT =/< 2.5 times the upper institutional limits of normal (=/<5 times the upper institutional limits of normal if hepatic metastases are present
* Adequate renal function as defined: by serum creatine =/< 1.5 times the upper limits of normal
* Adequate recovery from recent surgery, chemotherapy and radiation therapy. At least one week must have elapsed from the time of a minor surgery, at least 3 weeks for major surgery, chemotherapy and radiation therapy
* Life expectancy of at least 12 weeks
* ECOG performance status of 0-1
* At least 18 years old
* Willing and able to give written informed consent
* Accessible for treatment and follow-up. Patients enrolled in this trial must be treated at the participating center
* Women of Child Bearing Potential (WOCP) must have a negative serum or urine pregnancy test (minimum sensitivity IU/L or equivalent units of HCG) within 72 hours prior to start of study medication.

WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea=/>12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35mIU/mL]. Even women who are using oral, implanted or, injectable intrauterine device or barrier methods (diaphragm, condoms, spermicide) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential.

Exclusion Criteria

* More than one prior chemotherapy regimen for Stage IIIB or IV or for metastatic recurrent disease. Prior adjuvant or neoadjuvant chemotherapy is allowed.
* Patients who are candidates for curative resection.
* CTC Grade 2 or greater neuropathy (motor or sensory)
* Known brain metastases
* Prior radiation must have not included major bone marrow containing areas (pelvis, lumbar, spine) and must not have contained a target lesion as the only measurable lesion. A recovery period of at least 3 weeks after completion of radiotherapy is required prior to enrollment.
* Myocardial infarction, unstable angina, or any history of congestive heart failure within six months of study therapy
* Pregnant or breast-feeding women, or sexually active women of childbearing potential not using an adequate method of birth control.
* Sexually active fertile men, whose partners are women of childbearing potential, unless using an adequate method of birth control
* Serious intercurrent infections, or nonmalignant medical illnesses that are controlled or whose control may be jeopardized by the complications of this therapy
* Psychiatric disorders or other conditions rendering the patient incapable of complying with the requirements of the the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Un of California Davis Cancer Center, Sacramento, California
  - Mount Sinai Medical Center, Miami Beach, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Rush Presbyterian St Lukes ME, Chicago, Illinois
  - Consultants in Blood Disorders, Louisville, Kentucky
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - University of Maryland Greenbaum Cancer Center, Baltimore, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - University of Missouri/Ellis Fischel Cancer Center, Columbia, Missouri
  - Dartmouth-Hitchcock /Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Unviversity of North Carolina, Chapel Hill, North Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Vanderbilt University Med School Div of Medical Oncology, Nashville, Tennessee
  - University of Wisconsin Hospital, Madison, Wisconsin

REFERENCES:
- [Background] Vansteenkiste J, Lara PN Jr, Le Chevalier T, Breton JL, Bonomi P, Sandler AB, Socinski MA, Delbaldo C, McHenry B, Lebwohl D, Peck R, Edelman MJ. Phase II clinical trial of the epothilone B analog, ixabepilone, in patients with non small-cell lung cancer whose tumors have failed first-line platinum-based chemotherapy. J Clin Oncol. 2007 Aug 10;25(23):3448-55. doi: 10.1200/JCO.2006.09.7097. Epub 2007 Jul 2. PMID 17606973